CLINICAL TRIAL: NCT06933355
Title: Acute Effects of SGLT2 Inhibitor on Kidney Allograft Oxygen Tension: A Randomized, Double-blind, Placebo Controlled Crossover Trial
Brief Title: Acute Effects of SGLT2 Inhibitor on Kidney Allograft Oxygen Tension
Acronym: SGL-TX-MR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT:2024-513765-40-00
Record Dates: First submitted 2025-04-01; First posted 2025-04-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation Recipients; Magnetic Resonance Imaging (MRI); Sodium-Glucose Transporter 2 Inhibitors; Non-Diabetic Patients; Randomized Controlled Trial; Placebo Control Design
Keywords: SGLT2i; Kidney Transplant; Kidney Transplant Recipients; MRI; Magnetic resonance Imaging; BOLD-MRI; Blood oxygen level dependent MRI; non-diabetic patients; Sodium-glucose Transporter 2 inhibitors; RCT
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, placebo controlled, cross-over intervention study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT2i (Active Comparator): Single dose of SGLT2i (Jardiance 50 mg)
  Interventions: Drug: JARDIANCE 25mg
- Placebo (Placebo Comparator): Single dose placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JARDIANCE 25mg — The intervention will be SGLT2i compared with placebo. The trial include a total of 8 non-diabetic kidney transplant recipients.
  4 patients will randomly be assigned to start in the active arm, and treated with a single dose SGLT2i at intervention day 1 and a single dose placebo at intervention day 2.
  4 patients will randomly be assigned to start in the non-active arm, each participant will be treated with a single dose placebo at intervention day 1 and a single dose SGLT2i at intervention day 2.
  Other Names: SGLT2i
  Arms: SGLT2i
Drug: Placebo — The intervention will be SGLT2i compared with placebo. The trial include a total of 8 non-diabetic kidney transplant recipients. 4 patients will randomly be assigned to start in the active arm, and treated with a single dose SGLT2i at intervention day 1 and a single dose placebo at intervention day 2. 4 patients will randomly be assigned to start in the non-active arm, each participant will be treated with a single dose placebo at intervention day 1 and a single dose SGLT2i at intervention day 2.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate if a single dose of oral SGLT2i, (50 mg Jardiance) will change oxygen tension in the kidney transplant.

The main questions it aims to answer are:

* Does a single dose of oral SGLT2i (50 mg Jardiance) change oxygen tension in the kidney transplant cortex and medulla, estimated by magnetic resonance imaging?
* Does a single dose of oral SGLT2i (50 mg Jardiance) change kidney transplant cortical and medullary perfusion?
* Does a single dose of oral SGLT2i (50 mg Jardiance) change kidney transplant artery blood flow?
* Does a single dose of oral SGLT2i (50 mg Jardiance) change blood glucoses, blood pressure and heart rate?

Researchers will compare a single dose of oral SGLT2i (50 mg Jardiance) to a placebo (a look-alike substance that contains no drug) to see if a single dose of oral SGLT2i (50 mg Jardiance) changes oxygen tension in the kidney transplant.

Kidney transplant recipients with out diabetes will:

* Meet for two intervention days.
* A single dose of oral SGLT2i (50 mg Jardiance) or placebo will be given in random order, separated by at least 2 week washout period, the experiment will be repeated with the opposite treatment.
* Kidney cortex oxygenation, and blood flow in different compartments of the kidney transplant, is estimated by blood-oxygen-dependent level magnetic resonance imaging (BOLD-MRI). Patients are evaluated by routine clinical examination and routine biochemical measures for kidney transplant patients.

DETAILED DESCRIPTION:
Background:

Kidney transplantation is the best treatment of end-stage renal disease (ESRD), although median allograft survival is only 15 years. In non-transplant diabetic and non-diabetic patient's sodium-glucose co-transporter type 2 inhibitors (SGLT2i) protect kidney function, possibly by reducing the proximal tubule transport workload with subsequent improvement of renal oxygenation and relieve hypoxia.

Hypothesis:

SGLT2i in kidney transplant recipients (KTR) will improve kidney allograft cortex oxygenation.

Research Objective:

We aim to test the acute effect of SGLT2i on kidney allograft oxygen tension.

Design:

A randomized, double-blind, placebo-controlled, crossover intervention study. Designed according to the CONSORT statement

Methods:

A single dose of oral SGLT2i (50 mg Jardiance) and placebo in random order, separated by at least 2 week washout period, the experiment will be repeated with the opposite treatment.

Kidney cortex oxygenation and blood flow in different compartments of the kidney allograft will be estimated by blood-oxygen-dependent level magnetic resonance imaging (BOLD-MRI). Patients will be evaluated by routine clinical examination and routine biochemical measures for transplant patients.

Primary endpoint:

- Kidney allograft cortical and medullary oxygen tension, estimated by BOLD-MRI based renal T2* relaxation rate.

Secondary endpoint:

* Renal cortical and medullary perfusion ml/100 g/min
* Renal artery blood flow ml/min
* Blood glucose mmol/L
* Systolic blood pressure (SysBP) and diastolic blood pressure (DiaBP) mmHg
* Heart rate (HR), beats min-1

Study population:

8 Non-diabetic kidney transplant recipients > 6 months post-transplant and stable eGFR >20 ml/min will be recruited from Odense University Hospital (OUH) kidney transplant outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥ 18 years.
* Non-diabetic kidney transplant recipients
* > 6 months post-transplant
* Stable eGFR> 20 ml/min (defined as eGFR 20 ml/min ± 5 ml/min variation in the last 3 months)
* Immunosuppressive: Tacrolimus (Adport) and Mycophenolatmofetil (Myfenax/Cellcept/Mycophenolatmofetil)
* Capable of lying in a MR-scanner
* Capable of providing a signed informed consent and comply with study requirements.

  * Negativ pregnancy test

Exclusion Criteria:

* Diabetic kidney disease type 1 or 2 (World Health Organization (WHO) criteria)

  * Hemoglobin A1c ≥ 48 mmol/mol
  * Fasting venous plasma glucose ≥ 7,0 mmol/l or
  * 2-hours venous plasma glucose ≥ 11,1 mmol/l after oral glucose tolerance test (OGTT).
* Renal allograft failure (eGFR< 20 ml/min)
* Alanine aminotransferase (ALAT) > 3 x upper normal limit
* Bilirubin > 2 x upper normal limit
* Prednisone treatment
* Pregnancy
* Breastfeeding
* Exclusion criteria for MRI o Claustrophobia/physical not able to lie in MR-s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Kidney allograft cortex oxygenation, T2* | T2* measured at baseline, 3 and 6 hours post-intervention
  BOLD-MRI, T2* cortex, s-1

SECONDARY OUTCOMES:
Renal cortical perfusion, (ml/100g/min) | Renal cortical perfusion, measured at baseline, 3 and 6 hours post-intervention
  BOLD-MRI estimated renal cortical perfusion, (ml/100 g/min)

OTHER OUTCOMES:
Renal allograft artery blood flow (ml/min) | Renal allograft artery blood flow measured at baseline, 3 and 6 hours post-intervention
  BOLD-MRI, renal allograft artery blood flow (ml/min)
Blood glucose (mmol/L) | Blood glucose, measured at baseline, 3 and 6 hours post-intervention
  Blood glucose (mmol/L), estimated by handheld blood glucose meter
Blood pressure | Bloodpressure measured at baseline, 3 and 6 hours post-intervention
  Systolic and diastolic blood pressure (mmHg), Estimated by a validated blood pressure device.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte B Lange, MD, Principal Investigator — Department of Nephrology, Odense University Hospital
Locations (1):
- Department of Nephrology, Odense University Hospital Kløvervænget 6, Enterance 93, 3. floor, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Statement:
  Data Available:
  Individual participant data (IPD) that underlie the results reported in the published article will be shared after de-identification. This includes text, tables, figures, and appendices.
  Supporting Documents:
  The study protocol and statistical analysis plan will also be made available.
  Time Frame:
  Data will be shared immediately following publication. There is no specified end date for availability.
  Criteria for Access:
  Data will be shared with researchers who submit a methodologically sound proposal aimed at achieving the goals outlined in their approved research proposal.
  Access Mechanism:
  Interested researchers should direct their proposals to: lotte.borg.lange@rsyd.dk.
  To gain access, requestors will be required to sign a data access agreement.
  Data Storage:
  The data will be stored for 25 years on a secure third-party platform (OPEN).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available after the last patients last visit, which is estimated for summer 2025
  Data Storage:
  The data will be stored for 25 years on a secure third-party platform (OPEN).
Access Criteria: Criteria for Access:
  Data will be shared with researchers who submit a methodologically sound proposal aimed at achieving the goals outlined in their approved research proposal.
  Access Mechanism:
  Interested researchers should direct their proposals to: lotte.borg.lange@rsyd.dk.
  To gain access, requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Lange LB, Bistrup C. SGL-TX-MR-study protocol acute effects of SGLT2 inhibitor on kidney allograft oxygen tension, a randomized, double-blind, placebo controlled crossover trial. Trials. 2025 Dec 29;26(1):585. doi: 10.1186/s13063-025-09244-4. PMID 41462489